CLINICAL TRIAL: NCT02481518
Title: Preloading Magnesium Attenuate Cisplatin-induced Nephrotoxicity
Acronym: PRAGMATIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2558/172
Record Dates: First submitted 2015-05-17; First posted 2015-06-25 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Kidney Injury
Keywords: Cisplatin nephrotoxicity; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium (Experimental): Magnesium preloading group : Magnesium preloading for Cisplatin treatment
  Interventions: Drug: Magnesium
- Control (Active Comparator): Control group : Normal saline preloading for cisplatin treatment
  Interventions: Other: Control

INTERVENTIONS:
Drug: Magnesium — Pre loading fluid with Magnesium sulphate 16 milliequivalent plus potassium chloride 20 milliequivalent in Normal saline 500 ml IV drip in 4 hours before Cisplatin administration
  Arms: Magnesium
Other: Control — Potassium chloride 20 milliequivalent in Normal saline 500 ml IV drip in 4 hours before Cisplatin administration
  Other Names: Normal saline
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether magnesium preloading reduce incident of cisplatin induced acute kidney injury in head and neck cancer who receiving low dose cisplatin (40 mg/m2 weekly for 7 weeks).

DETAILED DESCRIPTION:
Randomized controlled trial comparing efficacy of magnesium preloading versus normal saline for prevention of acute and chronic nephrotoxicity of cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Eastern Cooperative Oncology Group score 0-2
* First Diagnosed Head and neck cancer and plan for treatment with cisplatin
* Serum creatinine ≤1.5 mg/dl or eGFR≥60(ml/min/1.73 m2)

Exclusion Criteria:

* Prior treatment with cisplatin before randomization
* Uncontrolled concurrent disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 7 days after cisplatin administration
  Comparing serum creatinine before Cisplatin treatment and seven days after cisplatin treatment

SECONDARY OUTCOMES:
Nephrotoxicity | up to 12 weeks
  Compare serum creatinine before Cisplatin treatment and complete 7 cycles of cisplatin treatment ( up to 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Arkom Nongnuch, MD, Principal Investigator — Ramathibodi hospital, Mahidol university
Locations (1):
- Faculty of medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand